CLINICAL TRIAL: NCT03875573
Title: Neo-adjuvant Chemotherapy Combined With Stereotactic Body Radiotherapy to the Primary Tumour +/- Durvalumab, +/- Oleclumab in Luminal B Breast Cancer: a Phase ll Randomised Trial
Brief Title: Neo-adjuvant Chemotherapy Combined With Stereotactic Body Radiotherapy to the Primary Tumour +/- Durvalumab, +/- Oleclumab in Luminal B Breast Cancer:
Acronym: Neo-CheckRay
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Institut Curie (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IJB-LBC-NEOCHECKRAY-2018
Record Dates: First submitted 2019-02-08; First posted 2019-03-14 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-03

CONDITIONS: Luminal B
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — durvalumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Neo-CheckRay is a multicenter, open-label phase II study that randomizes luminal B breast cancer subjects candidate for neo-adjuvant chemotherapy in a 1:1:1 ratio in 3 arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Chemotherapy and radiotherapy (Experimental): The combination of weekly paclitaxel 80 mg/m² IV followed by q2w dose-dense doxorubicin-cyclophosphamide (ddAC) (60 mg/m² doxorubicin IV and 600 mg/m² cyclophosphamide IV) and pre-operative radiation therapy on the primary tumour (3x8 Gy).
  Interventions: Radiation: Stereotactic Body Radiotherapy
- Chemotherapy and pre-operative radiotherapy plus durvalumab (Experimental): The combination of weekly paclitaxel 80 mg/m² IV followed by q2w dose-dense doxorubicin-cyclophosphamide (ddAC) (60 mg/m² doxorubicin IV and 600 mg/m² cyclophosphamide IV) and pre-operative radiation therapy on the primary tumour (3x8 Gy) with the addition of the anti-PD-L1 antibody durvalumab IV 1500 mg q4w.
  Interventions: Drug: Durvalumab; Radiation: Stereotactic Body Radiotherapy
- Chemotherapy & pre-op radiotherapy + durvalumab + oleclumab (Experimental): The combination of weekly paclitaxel 80 mg/m² IV followed by q2w dose-dense doxorubicin-cyclophosphamide (ddAC) (60 mg/m² doxorubicin IV and 600 mg/m² cyclophosphamide IV) and pre-operative radiation therapy on the primary tumour (3x8 Gy) with the addition of the anti-PD-L1 antibody durvalumab IV 1500 mg q4w and the addition of the anti-CD73 antibody oleclumab IV 3000 mg q2w for 4 administrations, followed by q4w for 3 administrations.
  Interventions: Drug: Durvalumab; Radiation: Stereotactic Body Radiotherapy; Drug: Oleclumab

INTERVENTIONS:
Drug: Durvalumab — an anti PD-L1 intravenous administration at 1500 mg every 4 weeks for 19 weeks.
  Other Names: MEDI4736
  Arms: Chemotherapy & pre-op radiotherapy + durvalumab + oleclumab; Chemotherapy and pre-operative radiotherapy plus durvalumab
Radiation: Stereotactic Body Radiotherapy — Pre-operative radiation therapy (boost dose) 3x8 Gy on the primary tumour at week 5 given in 3 fractions. The 3 fractions will be spread at the minimum over 3 days and at the maximum over 6 days.
  Other Names: SBRT
Drug: Oleclumab — an anti-CD73 intravenous administration at 3000 mg every 2 weeks for the first 4 administrations then every 4 weeks for the last 3 administrations.
  Other Names: MEDI9447
  Arms: Chemotherapy & pre-op radiotherapy + durvalumab + oleclumab

SUMMARY:
Neo-CheckRay is a multicenter, open-label phase II study that randomizes luminal B breast cancer subjects candidate for neo-adjuvant chemotherapy in a 1:1:1 ratio in 3 arms:

1. the combination of weekly paclitaxel followed by dose-dense doxorubicin-cyclophosphamide (ddAC) and pre-operative radiation therapy (boost dose) on the primary tumour
2. arm 1 with the addition of the anti-PD-L1 antibody durvalumab
3. arm 2 with the addition of the anti-CD73 antibody oleclumab The primary tumour will be excised 2-6 weeks after completion of ddAC. A safety run-in is planned for the 6 first subjects before starting the randomized phase II trial. Those 6 subjects will receive the treatment given in Arm 3.

DETAILED DESCRIPTION:
This trial consists of a safety run-in followed by a phase II randomised trial. The goal of the safety run-in is to assess the safety of adding SBRT to the neo-adjuvant systemic treatment. The doses of the IMPs will be identical in the safety run-in and the phase II randomised trial. Individual subject timelines are also identical in the safety run-in and the phase II randomised trial.

The safety run-in is done as a precursor to the phase II randomised part of the Neo-CheckRay trial. Six subjects will be included in the safety run-in. These subjects are not part of the phase II total recruitment.

Subjects in the safety run-in will receive the following treatments corresponding to arm 3 of the phase II randomised trial. This consists of:

* q1w paclitaxel 80 mg/m² IV for 12 administration (12 weeks) followed by q2w dose-dense doxorubicin-cyclophosphamide IV (60 mg/m² and 600 mg/m² respectively) for 4 administrations (8 weeks)
* Anti-PD-L1 antibody durvalumab 1500 mg IV q4w for 5 administration (20 weeks)
* Anti-CD73 antibody oleclumab 3000 mg IV q2w for 4 administrations (8 weeks), followed by q4w for 3 administrations (12 weeks)
* Pre-operative radiation therapy (boost dose) 3x8 Gy on the primary tumour at week 5

If all requirements are meet during the safety run-in, then the phase II part of the study will be opened. The phase II will consist of luminal B breast cancer subjects candidate for neo-adjuvant chemotherapy will be randomised in a 1:1:1 ratio between 3 arms:

1. Arm 1: the combination of weekly paclitaxel 80 mg/m² IV followed by q2w dose- dense doxorubicin-cyclophosphamide (ddAC) (60 mg/m² doxorubicin IV and 600 mg/m² cyclophosphamide IV) and pre-operative radiation therapy on the primary tumour (3x8 Gy).
2. Arm 2: drugs regimen of Arm 1 with the addition of the anti-PD-L1 antibody durvalumab IV 1500 mg q4w.
3. Arm 3: drugs regimen of Arm 2 with the addition of the anti-CD73 antibody oleclumab IV 3000 mg q2w for 4 administrations, followed by q4w for 3 administrations.

The primary tumour will be excised 2-6 weeks after completion of ddAC. The study treatments end at surgery. All treatment after surgery, such as post-operative radiotherapy and hormonal therapy, will be performed according to standard of care and local site guidelines. The patient will then be followed for the next 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Female
* ECOG performance status ≤ 1
* Weight ≥ 35 kg
* Histological diagnosis of invasive breast adenocarcinoma that is estrogen receptor-positive (ER-positive) and HER2- negative, as per the updated American Society of Clinical Oncology (ASCO) - College of American Pathologists (CAP) guidelines and performed according to local testing. In addition, only tumours with Proliferation Index Ki67 ≥ 15% or histology grade III are accepted.
* Agreement to perform new study related biopsies to provide tissue samples
* MammaPrint genomic high risk score according to centralised testing, except for specific conditions as mentioned below. Mammaprint will only be tested for luminal B breast tumours with either Proliferation Index Ki67 ≥ 15% or histology grade III tumours. (Testing to be done during screening period).

MammaPrint result status at time of termination of all other screening procedures

* MammaPrint is high risk: subject may be randomized.
* MammaPrint is low risk: subjet can not be randomized.
* MammaPrint result is not yet known:

If the MammaPrint result is not known at time of termination of all other screening procedures, the investigator is allowed to randomize the subject and start study treatment without waiting for the result of the MammaPrint in the following situations: (Ki67 > 20 % or grade III) and Age<50 years+ cN0 OR Age ≥ 50 years + cN+ • Tumour size:

* If subject is cN0: tumour size ≥ 2 cm, as determined by MRI imaging.
* If subject is cN1, cN2 or cN3: tumour size ≥ 1.5 cm, as determined by MRI imaging.

The requirement for an MRI is not applicable in the case of medical contraindications to perform MRI (e.g., obesity or claustrophobia). In this situation, tumour evaluations should be performed by ultrasound.

* Multifocal, multicentric unilateral or bilateral breast adenocarcinoma tumours are allowed provided that all biopsiable foci are ER+/HER2- according to local testing and all foci are able to receive SBRT treatment within the defined dosimetric constraints. In some cases a separate biopsy of every focus is not mandatory, but only if every of the following conditions are present:

  -small focal lesion

  -lesion in close proximity to the main primary cancer from which a biopsy was taken
  * the investigator and the radiologist consider the lesion to be clearly related to the main primary breast cancer from which a biopsy was taken
  * the lesion will be removed during the same lumpectomy than the main primary breast cancer For bilateral, multifocal or multicentric disease, the site selected for pre-treatment biopsy should correspond to the site of largest measurable disease meeting eligibility criteria. The location of tumour biopsy site (laterality, quadrant, position from the nipple and type of imaging modality to guide biopsy) should be collected.
* Serum pregnancy test (for subjects of childbearing potential) negative within 2 weeks prior to first dose of study administration.
* Women of childbearing potential must agree to use 1 highly effective method of contraception during the screening period, during the course of the study and at least 12 months after the last administration of study treatment. it is strongly recommended for the male partner of a female subject to also use male condom plus spermicide throughout this period.
* Adequate bone marrow function as defined below:

  * Absolute neutrophil count ≥1500/µL, i.e. 1.5x10^9/L
  * Hemoglobin ≥ 9.0 g/dL
  * Platelets ≥100000/µL, i.e. 100x10^9/L
* Adequate liver function as defined below:

  - Serum total bilirubin ≤ 1.5 x ULN. In case of known Gilbert's syndrome ≤ 3 x UNL is allowed

  - AST (SGOT) ≤ 3.0 x ULN
  * ALT (SGPT) ≤ 3.0 x ULN
* Adequate renal function as defined below:

  * Creatinine ≤ 1.5 x UNL or eGFR ≥ 40ml/min/1.73m²
* Adequate coagulant function as defined below:

  * International Normalized Ratio (INR) ≤ 1.5 x ULN
* Completion of all necessary screening procedures within 28 days prior to randomisation (except if written differently).
* Willingness to provide tissue and blood samples for immuno-monitoring and translational research activities
* Left ventricular ejection fraction (LVEF) ≥ 50%. LVEF performed in routine is accepted if done within 6 months prior to beginning of screening.
* Signed Informed Consent form (ICF) obtained prior to any study related procedure.

Inclusion criterion for phase II only (all phase II subjects):

• Tumour sample provided for central PD-L1 IHC assessment. (Testing done during screening period).

Inclusion criterion applicable to FRANCE only (all safety run-in and phase II subject):

• Affiliated to the French Social Security System (applicable only to subjects treated in France)

Exclusion Criteria:

* Pregnant and/or lactating women.
* Subject with a significant medical, neuro-psychiatric, substance abuse or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.
* TNM stage cT4 breast cancer including inflammatory breast cancer
* Presence of any distant metastasis
* Contra-indication for treatment by paclitaxel, doxorubicin or cyclophosphamide, or known allergy to any tested substances or any excipients (e.g; chemotherapy or immunotherapy formulations). Contra-indication for subjects with known sensitivity to acetaminophen/paracetamol, diphenhydramine or equivalent antihistamine (this is a contra-indication for treatment with oleclumab).
* Previously known contra-indication for treatment by radiation therapy such as rare genetic disorders associated with DNA repair disorders such as ataxia-telangiectasia (A-T), Nijmegen Breakage Syndrome (NBS) and Fanconi anemia.
* Active or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, Wegner's granulomatosis) within the past 3 years. NOTE: Subjects with childhood atopy or asthma, vitiligo, alopecia, Grave's disease, Hashimoto's thyroiditis, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Prior malignancy active within the previous 5 years, except for localised cancers that are considered to have been cured and in the opinion of the investigator present a low risk for recurrence. Examples include basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast
* Known history of, or any evidence of active, non-infectious pneumonitis.
* Active infection including:

  * Tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice)
  * Hepatitis B (known positive HBV surface antigen (HBsAg) result). Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.
  * Hepatitis C. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction, transient ischemic attack, or stroke within the previous 3 months, unstable arrhythmias, and/or unstable angina
* Medical condition requiring current systemic anticoagulation, or a history of congenital hypercoagulable condition. Subjects taking aspirin at doses < 325 mg per day are eligible provided that prothrombin time is within the institutional range of normal. Use of local anticoagulation for port maintenance is permitted.
* Subjects with history of venous thrombosis in the past 12 months prior to the scheduled first dose of study treatment (oleclumab).
* Diabetes mellitus Type 1 or poorly controlled Type 2 diabetes mellitus defined as a screening hemoglobin A1C ≥ 8 % or a fasting plasma glucose ≥ 160 mg/dL (or 8.8 mmol/L)
* Any live (attenuated) vaccine within 30 days of planned start of study therapy.
* Prior systemic immunosuppressive medication (excluding corticosteroids) within 30 days of planned start of study therapy.
* Prior radiation therapy to the ipsilateral breast.
* Prior immunotherapy, including tumour vaccine, cytokine, anti-CTLA4, PD-1/PD-L1, including durvalumab, blockage or similar agents.
* Concomitant use of other investigational drugs
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria. Subjets with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician. Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or oleclumab may be included only after consultation with the Study Physician.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the subject to give written informed consent.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Prior organ transplantation
* Subjects with urinary outflow obstruction

Exclusion criterion applicable to FRANCE only

• Vulnerable persons according to the article L.1121-6 of the CSP, adults who are the subject of a measure of legal protection or unable to express their consent according to article L.1121-8 of the CSP.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be female by biological birth.
Enrollment: 147 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety Run-in: Evaluation of the immune related or radiation therapy related toxicity of special interest | 7 months
  Immune related or radiation therapy related toxicity of special interest are identifitied as:
  * Any Grade 4 immune-related AE
  * Any ≥ Grade 3 colitis
  * Any ≥ Grade 3 renal failure/nephritis
  * Any ≥ Grade 3 non-infectious pneumonitis irrespective of duration
  * Any Grade 3 immune-related AE, excluding colitis, renal failure/nephritis and pneumonitis, that does not downgrade to ≤ Grade 2 within 3 days after onset of the event despite maximal medical supportive care including systemic corticosteroids or does not downgrade to ≤ Grade 1 or baseline within 14 days
  * Liver transaminase elevation ≥ 5 ULN or total bilirubin > 3 × ULN will be considered a DLT regardless of duration or reversibility
  * Any increase in AST or ALT > 3 × ULN and concurrent increase in total bilirubin > 2 × ULN
Safety Run-in: Evaluation of the feasibility of the primary surgery | 7 months
  Feasibility of performing surgery within 6 weeks after the last neo-adjuvant treatment. This would indicate that there were no significant delays or toxicities that would results in surgery being delayed.
Phase II: Demonstration of the tumour response in arms 2 or 3 versus arm 1 | 24 months
  To demonstrate improved tumour response of the primary tumour and nodal metastases in arms 2 or 3 versus arm 1 using residual cancer burden (RCB 0-1 vs. RCB 2-3) at time of surgery.

SECONDARY OUTCOMES:
Phase II: Evaluation of the rthe complete pathological response rate defined as ypT0/Tis ypN0 | 24 months
  Absence of residual invasive disease, residual in situ carcinoma is accepted.
Phase II: Evaluation of the complete pathological response rate defined as ypT0 ypN0 | 24 months
  absence of residual invasive disease and in situ carcinoma.
Phase II: Evaluation of the response to the primary tumour irrespective of the response to the pathological lymph nodes | 24 months
  Complete pathologic response rate (pCR) of the primary tumour (ypT0/ Tis), irrespective of the response rate of the resected nodal metastases
Phase II: Evaluation of the response to the pathological lymph nodes irrespective of the response to the primary tumour | 24 months
  Complete pathologic response rate (pCR) of the resected nodal metastases (ypN0), irrespective of the response rate of the primary tumour.
Phase II: Evaluation of the the feasibility to perform breast-sparing surgery of the arms 2 and 3 versus arm 1 | 24 months
  % of breast conservation surgery in arms 2 and 3 versus arm 1
Phase II: Demonstration of the an increase in TIL levels of the primary breast cancer between baseline and the week 6 biopsy | 24 months
  Change in TIL levels between baseline and the week 6 biopsy.
Phase II: Evaluation of the ability to control invasive disease and survival in arms 2 and 3 versus arm 1 at year 3 and 5 years after surgery | 5 years
  Efficacy endpoints at 3 years and 5 years after surgery will be measured, as defined by the Standardized Definitions for Efficacy End Points in Neoadjuvant Breast Cancer Clinical Trials (NeoSTEEP) (88). The following endpoints will be assessed: event-free survival (EFS), breast cancer event-free survival (BC-EFS), overall survival (OS) and distant recurrence-free survival (DRFS). Furthermore, the occurrence of ipsilateral locoregional recurrence (breast, chestwall or locoregional nodal recurrence), ipsilateral local recurrence (breast or chest wall) (laterality of the index lesion), and ipsilateral locoregional nodal recurrence (laterality of the index lesion) will be assessed. The endpoints will be measured using regular follow-up investigations: lab work, clinical examination and annual breast ultrasound and mammography. Radiologic imaging will not be routinely performed, unless directed by abnormal blood results or clinical examination.
Phase II: Evaluation of the severity and duration of AEs of the arms 2 and 3 versus arm 1 | 5 years
  Duration and severity of AEs based on CTCAE 5.0
Phase II: Evaluation of the the cosmetic changes to the breast of the arms 2 and 3 versus arm 1 | 5 years
  Changes in breast appearance: breast fibrosis in whole breast, breast fibrosis in boost area, breast size, breast shape, nipple position, shape of the areola and nipple, skin color, appearance of surgical scar, evaluation of teleangiectasia and global cosmetic result. Information on cosmetic and plastic surgical procedures will be collected (for example: oncoloplastic surgery, breast implants, and other procedures).

CONTACTS AND LOCATIONS:
Overall Officials: Alex De Caluwe, MD, Study Chair — Jules Bordet Institute
Locations (7):
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitaire Ziekenhuizen, Leuven
  - CHU UCL Namur Sainte-Elisabeth, Namur
  - GZA - Ziekenhuizen (Campus St. Augustinus), Wilrijk
- France (2):
  - Centre Georges François Leclerc, Dijon
  - Institut Curie, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Caluwe A, Romano E, Poortmans P, Gombos A, Agostinetto E, Marta GN, Denis Z, Drisis S, Vandekerkhove C, Desmet A, Philippson C, Craciun L, Veys I, Larsimont D, Paesmans M, Van Gestel D, Salgado R, Sotiriou C, Piccart-Gebhart M, Ignatiadis M, Buisseret L. First-in-human study of SBRT and adenosine pathway blockade to potentiate the benefit of immunochemotherapy in early-stage luminal B breast cancer: results of the safety run-in phase of the Neo-CheckRay trial. J Immunother Cancer. 2023 Dec 6;11(12):e007279. doi: 10.1136/jitc-2023-007279. PMID 38056900
- [Derived] De Caluwe A, Buisseret L, Poortmans P, Van Gestel D, Salgado R, Sotiriou C, Larsimont D, Paesmans M, Craciun L, Stylianos D, Vandekerckhove C, Reyal F, Isabelle V, Eiger D, Piccart M, Romano E, Ignatiadis M. Neo-CheckRay: radiation therapy and adenosine pathway blockade to increase benefit of immuno-chemotherapy in early stage luminal B breast cancer, a randomized phase II trial. BMC Cancer. 2021 Aug 6;21(1):899. doi: 10.1186/s12885-021-08601-1. PMID 34362344